CLINICAL TRIAL: NCT03015350
Title: Blood Levels of Sevoflurane and Desflurane During One Lung Ventilation
Brief Title: Blood Levels of Sevoflurane and Desflurane
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, MD, Anesthesiology specialist, Cukurova University
Other Study IDs: One lung ventilation
Record Dates: First submitted 2016-12-27; First posted 2017-01-10 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2017-11

CONDITIONS: Anesthetics, Inhalation
Keywords: blood sevoflurane concentration; blood desflurane concentration; one lung ventilation
MeSH Terms: conditions — Respiratory Aspiration | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- two lung ventilation of Sevoflurane: In GroupSa, 1,5 % sevoflurane will be apply continuously and blood samples will be taken at intervals of 10 minutes starting from the 40th minute.
  Interventions: Drug: Sevoflurane
- one lung ventilation of Sevoflurane: In GroupSa, 1,5 % sevoflurane will be apply continuously and first samples will taken at the 40. minutes and collection of blood samples will be continue at intervals of 10 minutes after one lung ventilation started.
  Interventions: Drug: Sevoflurane
- two lung ventilation of Desflurane: In GroupSa, 6 % desflurane will be apply continuously and blood samples will be taken at intervals of 10 minutes starting from the 40th minute.
  Interventions: Drug: Desflurane
- one lung ventilation of desflurane: In GroupSa, 6 % desflurane will be apply continuously and first samples will taken at the 40. minutes and collection of blood samples will be continue at intervals of 10 minutes after one lung ventilation started.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Measurement of blood desflurane level during one lung ventilation
  Other Names: Blood sevoflurane level
  Groups: one lung ventilation of Sevoflurane; two lung ventilation of Sevoflurane
Drug: Desflurane — Measurement of blood desflurane level during one lung ventilation
  Other Names: Blood desflurane level
  Groups: one lung ventilation of desflurane; two lung ventilation of Desflurane

SUMMARY:
16 patients with American Society of AnesthesioIogy (ASA) physical status I-III will recruited to this study. Patients will divided to the 2 groups. %1.5 Sevoflurane will apply in Group S and %6 Desflurane will apply in Group D. Each groups will divide 2 subgroups. Two lung ventilation will be performed to Group Sa and Group Da, one lung ventilation will be performed to Group Sb and Group Db. At the time point 40.minutes first blood sample will given from patients. Blood sample will be taken at intervals of 10 minutes from groups of two lung ventilation. In groups of one lung ventilation, blood samples will be taken at the time interval of 10 minutes after one lung ventilation started. All blood samples will be assess in Gas Chromatography.

DETAILED DESCRIPTION:
Investigator aimed to assess blood level of sevoflurane and desflurane during two lung ventilation and one lung ventilation. The investigators will use Gas Chromatography for define drugs levels. 16 patients with ASA I-III patients who undergo thoracotomy and abdominal surgery will be recruited to this study. Patients will divided in to the 2 groups. %1.5 Sevoflurane will apply in Group S and %6 Desflurane will apply in Group D during anesthesia maintenance. Each groups will divide 2 subgroups which are one lung ventilation groups and two lung ventilation groups. Two lung ventilation will be performed to Group Sa and Group Da, one lung ventilation will be performed to Group Sb and Group Db. Sequential blood samples will be taken from both arterial and central venous canula at the same time point. First blood samples will be taken at 40. minutes of anesthesia. Sequential samples will be taken at interval of 10 minutes during two lung ventilation. In one lung ventilation second blood samples will be taken at the 10. minutes of one lung ventilation. After than at the interval of 10 minutes, collection of blood samples both arterial and central venous will be continue.

All collection will assess with gas chromatography.

ELIGIBILITY:
Inclusion Criteria: ASA I-II patients

* Who undergo thoracotomy or abdominal surgery

Exclusion Criteria:

* ASA IV and up patients
* Patients who taken inotropic agent

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 patients with ASA I-III who undergo thoracotomy or abdominal surgery
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Measurement of blood levels of Sevoflurane and Desflurane | from 40th minute to the end of the operation
  Data collections will be ensured from arterial and venous blood sample and than samples will be assessed with gas chromatography and blood sevoflurane and desflurane level will be measured. Blood samples will take every 10 minutes. Only blood levels of sevoflurane and desflurane will be assessed.

SECONDARY OUTCOMES:
determine of ventilation-perfusion mismatch with p(A-a)O2 | from 40th minute to the end of the one lung ventilation
  During one lung ventilation, p(a-A)O2 will be assessed with arterial blood analyses

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Biricik, MD, Principal Investigator — Cukurova University
Locations (1):
- Ebru Biricik, Adana, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No